CLINICAL TRIAL: NCT06062953
Title: Efficacy of Melatonin, Low-dose Quetiapine, or Placebo in Patients With Psychiatric Disorders and Comorbid Insomnia: a Randomized Clinical Trial
Brief Title: Efficacy of Melatonin, Low-dose Quetiapine, or Placebo in Patients With Psychiatric Disorders and Comorbid Insomnia
Acronym: MEL-QUE
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Lone Baandrup (Other)
Collaborators: Danish Center for Sleep Medicine (Other); Region Capital Denmark (Other); Copenhagen Trial Unit, Center for Clinical Intervention Research (Other); Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Responsible Party: Sponsor-Investigator, Lone Baandrup, Sponsor-investigator, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023-504728-24-00
Record Dates: First submitted 2023-09-13; First posted 2023-10-02 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Psychiatric Disorders; Insomnia
MeSH Terms: conditions — Mental Disorders; Sleep Initiation and Maintenance Disorders | interventions — Melatonin; Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Melatonin (Experimental)
  Interventions: Drug: Melatonin
- Quetiapine (Experimental)
  Interventions: Drug: Quetiapine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Melatonin — 3-9 mg flexible dosing before bed time
  Arms: Melatonin
Drug: Quetiapine — 50-150 mg flexible dosing before bed time
  Arms: Quetiapine
Drug: Placebo — 1-3 capsules flexible dosing before bed time
  Arms: Placebo

SUMMARY:
The goal of this investigator-initiated, randomized, blinded, 3-armed placebo-controlled, pragmatic, clinical superiority trial is to examine the efficacy of melatonin or low-dose quetiapine versus placebo for treatment of insomnia in patients with psychiatric disorders. The aims of the study are:

* To examine the efficacy of melatonin or low-dose quetiapine versus placebo for treatment of insomnia
* To examine how melatonin or low-dose quetiapine affects global symptom severity, sleep quality, psychosocial functioning and subjective well-being.

Participants will receive six weeks of treatment with either melatonin, quetiapine or placebo followed by a brief taper off.

ELIGIBILITY:
Inclusion Criteria:

* 16 to 64 years of age
* ICD-10 diagnosis of a current or previous mental or behavioral disorder (F20-F69, F84, F90-95)
* For the diagnoses F84 and F90 a previous period of treatment with melatonin is required
* For the 16-17 years old: Non-pharmacological treatment options including sleep hygiene education, weighted blanket or other gravity products have been tested with insufficient effect
* Self-reported sleep difficulties at least three times per week in the preceding 3 months
* Insomnia Severity Index score ≥11
* Women of childbearing potential: negative pregnancy test at baseline and use of highly effective contraception measures
* Informed consent

Exclusion Criteria:

* Current treatment with melatonin or quetiapine
* Severe somatic comorbidity
* BMI ≥ 35 kg/m2
* Breastfeeding
* Alcohol and/or substance dependency within the last 3 months
* Inadequate Danish language skills
* Not able to make an informed consent
* Increased cardiac risk as assessed by presence of cardiac risk factors, cardiac symptoms, or prolonged QT-interval at baseline ECG

Ages: 16 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 255 (Estimated)
Dates: Start 2023-09-18 (Actual); Primary Completion 2029-02-28 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Insomnia severity | 6 weeks
  Insomnia Severity Index, range 0-28, higher is worse

SECONDARY OUTCOMES:
Clinical global impression (CGI) | 6 weeks
  Clinical global impression: Severity, range 0-7, higher is worse
Subjective sleep quality | 6 weeks
  Pittsburgh Sleep Quality Index, range 0-21, higher is worse
Psychosocial functioning | 6 weeks
  Personal and Social Performance Scale, range 1-100, higher is better
Patient-reported subjective well-being | 6 weeks
  WHO-5 well-being index, range 0-100, higher is better

OTHER OUTCOMES:
Objective sleep quality (polysomnography) | 6 weeks
  Total sleep time in minutes, higher is better
Circadian rhythmicity (actigraphy) | 6 weeks
  Interdaily stability which quantifies the invariability from day to day, i.e., the predictability of the 24 h rest-activity pattern. This index will be 1 for perfect interdaily stability and thus lower values reflect higher variability between the observed days

CONTACTS AND LOCATIONS:
Overall Officials: Lone Baandrup, MD, Principal Investigator — Mental Health Center Copenhagen
Locations (1):
- Mental Health Center Copenhagen, Copenhagen NV, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be available for meta-analysis. Proposals should be directed to: lone.baandrup@regionh.dk. To gain access, data requestors will need to sign a data access agreement.
Supporting Information: Study Protocol, SAP
Time Frame: After publication of planned primary, secondary and exploratory outcomes. There will be no end date for availability of data.
Access Criteria: Meta-analytical purposes